CLINICAL TRIAL: NCT00564720
Title: Phase II Study of Gemcitabine Plus Erlotinib Versus Erlotinib Plus Gemcitabine Plus Oxaliplatin, in Patients With Locally Advanced or Metastatic Pancreatic Cancer
Brief Title: Gemcitabine Plus Erlotinib Versus Erlotinib Plus Gemcitabine Plus Oxaliplatin, in Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to poor accrual of the study
Sponsor: Hellenic Oncology Research Group (Other)
Collaborators: University Hospital of Crete (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT/06.13
Record Dates: First submitted 2007-11-27; First posted 2007-11-28 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Erlotinib Hydrochloride; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): GEM/TAR
  Interventions: Drug: Gemcitabine; Drug: Erlotinib
- 2 (Experimental): GEM/OX/TAR
  Interventions: Drug: Gemcitabine; Drug: Erlotinib; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine 1000mg/m2 IV on days 1, 8, and 15 every 28 days for 6 cycles
  Other Names: Gemzar
  Arms: 1
Drug: Gemcitabine — Gemcitabine 1100 mg/m2 IV on days 1 and 8 every 21 days for 6 cycles
  Other Names: Gemzar
  Arms: 2
Drug: Erlotinib — Erlotinib 100 mg by mouth (p.o.), daily until disease progression
  Other Names: Tarceva
Drug: Oxaliplatin — Oxaliplatin 130 mg/m2 IV on day 8, every 21 days for 6 cycles
  Other Names: Eloxatin
  Arms: 2

SUMMARY:
This randomized phase II trial will compare the efficacy and toxicity of Gemcitabine plus Erlotinib versus Gemcitabine plus Erlotinib plus Oxaliplatin in patients with pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed pancreatic cancer.
* Measurable disease.
* Absence of ascites or obstructive jaundice.
* ECOG Performance Status 0-2.
* Adequate liver kidney and bone marrow function.
* Written informed consent.

Exclusion Criteria:

* Chronic diarrheic syndrome.
* Uncontrolled brain metastases after radiation.
* Liver infiltration over 50%.
* Peripheral neuropathy ≥ 2.
* No second primary malignancy within the past 5 years, except non-melanomas skin cancer or in situ carcinoma of the cervix.
* No active uncontrolled infection.
* Active cardiac disease : unstable angina or onset of angina within last 3 months, myocardial infarction within 6 months, congestive heart failure > class II, cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
* Women who are pregnant or lactating.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2006-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 1 year survival

SECONDARY OUTCOMES:
Progression free interval | 1 year
Response rate | Objective responses confirmed by CT or MRI on 3rd and 6th cycle
Toxicity profile | Toxicity assessment on each chemotherapy cycle
Symptoms improvement | Assessment every two cycles

CONTACTS AND LOCATIONS:
Overall Officials: Vassilis Georgoulias, MD, Principal Investigator — University Hospital of Crete, Dep of Medical Oncology
Locations (8):
- Greece (8):
  - University General Hospital of Alexandroupolis, Department of Medical Oncology, Alexandroupoli
  - Air Forces Military Hospital of Athens, Athens
  - Errikos Ntynan General Hospital, Athens
  - IASO General Hospital of Athens, 1st Department of Medical Oncology, Athens
  - Laikon General Hospital, Medical Oncology Unit, Propedeutic Department of Internal Medicine, Athens
  - Metaxa's Anticancer Hospital of Piraeus, 1st Department of Medical Oncology, Athens
  - State General Hospital of Larissa, Larissa
  - Diabalkaniko General Hospital of Thessaloniki, Thessaloniki